CLINICAL TRIAL: NCT05828732
Title: Clinical Feasibility of Disease-managing Mobile Application in the Patients With Hyperthyroidism
Brief Title: Clinical Feasibility of Disease Managing Mobile App for Hyperthyroidism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: THYROSCOPE INC. (Industry)
Responsible Party: Principal Investigator, Jae Hoon Moon, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B-2201-735-304
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- app user group (Experimental): The participants in this group start using wearable devices to monitor their heart rate and a mobile app to assist with the management of hyperthyroidism after being diagnosed and beginning treatment with anti-thyroid medication.
  Interventions: Other: Using a mobile app that integrates with wearable devices
- non-user group (No Intervention): The participants in this group begin treatment with anti-thyroid medication after being diagnosed with thyrotoxicosis, but they do not use the wearable devices or mobile app used in this study.

INTERVENTIONS:
Other: Using a mobile app that integrates with wearable devices — Using a mobile app that integrates with wearable devices to monitor heart rate, check self-reported symptoms, provide disease-related information, and set medication reminders for patients with thyrotoxicosis.
  Arms: app user group

SUMMARY:
This randomized controlled study aims to investigate the effects of using a mobile app that integrates with wearable devices to monitor heart rate, check self-reported symptoms, provide disease-related information, and set medication reminders for patients with thyrotoxicosis. The study intends to evaluate how the use of the app affects disease progression, quality of life, and health-related behaviors associated with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been newly diagnosed or are currently undergoing treatment for thyrotoxicosis at Bundang Seoul National University Hospital.
* Subjects must be able to use the smartphone app required for the use of wearable devices and their integration.

Exclusion Criteria:

* Subjects who have constraints on normal activity due to diseases other than thyroid dysfunction.
* Subjects who are currently taking medication that affects heart rate.
* Subjects with heart conditions such as arrhythmia that affect heart rate.
* Subjects who cannot undergo antithyroid drug treatment and require surgery or radioactive iodine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Scores of quality of life assessed by SF-36 survey | baseline (at enrollment)
  Scores of quality of life assessed by SF-36 survey
Scores of quality of life assessed by SF-36 survey | 6 weeks after baseline
  Scores of quality of life assessed by SF-36 survey
Scores of quality of life assessed by SF-36 survey | 10 weeks after baseline
  Scores of quality of life assessed by SF-36 survey
Scores of quality of life assessed by SF-36 survey | 14 weeks after baseline
  Scores of quality of life assessed by SF-36 survey
antithyroidal drug compliance | 6 weeks after baseline
  Medication adherence assessed by directly counting the remaining pills after taking the prescribed medication.
antithyroidal drug compliance | 10 weeks after baseline
  Medication adherence assessed by directly counting the remaining pills after taking the prescribed medication.
antithyroidal drug compliance | 14 weeks after baseline
  Medication adherence assessed by directly counting the remaining pills after taking the prescribed medication.
Knowledge about hyperthyroidism | 14 weeks after baseline
  A score measured through a test designed to assess the knowledge level about Graves' disease

SECONDARY OUTCOMES:
free T4 | baseline
  serum free T4 concentration
free T4 | 6 weeks after baseline
  serum free T4 concentration
free T4 | 10 weeks after baseline
  serum free T4 concentration
free T4 | 14 weeks after baseline
  serum free T4 concentration
free T3 | baseline
  serum free T3 concentration
free T3 | 6 weeks after baseline
  serum free T3 concentration
free T3 | 10 weeks after baseline
  serum free T3 concentration
free T3 | 14 weeks after baseline
  serum free T3 concentration
TSH | baseline
  serum free TSH concentration
TSH | 6 weeks after baseline
  serum free TSH concentration
TSH | 10 weeks after baseline
  serum free TSH concentration
TSH | 14 weeks after baseline
  serum free TSH concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea